CLINICAL TRIAL: NCT05091099
Title: The Optimal Sequential Therapy After Long Term Denosumab Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202108044MINA
Record Dates: First submitted 2021-10-11; First posted 2021-10-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; denosumab; alendronate; zoledronic acid
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid; Alendronate

STUDY DESIGN:
Intervention Model Description: One arm accept on time zoledronic acid after long-tearm denosumab. Another arm accept alendronate for 4 months and then zoledronic acid after long-tearm denosumab.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On time Zoledronate (Active Comparator): Zoledronate would be given (one dose for one year) after the completiong of denosumab on time
  Interventions: Drug: zoledronate
- Alendronate and Zoledronate (Experimental): Alendronate would be given one month before the the completiong of denosumab and the following 3 months (Total four months). After the completion of Alendronate, Zoledronate would be given (one dose).
  Interventions: Drug: Alendronate and Zoledronate

INTERVENTIONS:
Drug: zoledronate — On time Zoledronate: Zoledronate would be given (one dose for one year) after the completiong of denosumab on time
  Other Names: Zoledronic acid
  Arms: On time Zoledronate
Drug: Alendronate and Zoledronate — Alendronate and Zoledronate: Alendronate would be given one month before the the completiong of denosumab and the following 3 months (Total four months). After the completion of Alendronate, Zoledronate would be given (one dose).
  Arms: Alendronate and Zoledronate

SUMMARY:
This study intends to investigate whether Alendronate and Zoledronate can prevent bone mineral density loss after long-term treatment with Denosumab.

DETAILED DESCRIPTION:
This study intends to use a randomized trial to test whether Alendronate and Zoledronate can avoid the risk of rapid bone loss after the withdrawal of Denosumab.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women or men over 50 years old
2. Continuous Denosumab treatment for at least three years (up to six doses).

Exclusion Criteria:

1. Secondary osteoporosis
2. Metabolic bone diseases
3. Active or prior malignancy
4. Ongoing systemic glucocorticoid therapy
5. Current use of hormone replacement therapy
6. Current use of any medication known to affect bone metabolism
7. Prior use of any osteoporosis medication other than denosumab
8. Estimated glomerular filtration rate (eGFR) < 40 mL/min
9. Known hypersensitivity to zoledronic acid
10. Hypocalcemia
11. Any other contraindication to zoledronic acid
12. Age > 85 years
13. Esophageal abnormalities that delay esophageal emptying (e.g., esophageal stricture, achalasia)
14. Inability to stand or sit upright for at least 30 minutes

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Bone mineral density of lumbar spine | one year
  Bone mineral density of lumbar spine

SECONDARY OUTCOMES:
Bone mineral density of femoral neck | one year
  Bone mineral density of femoral neck
Bone mineral density of total hip | one year
  Bone mineral density of total hip
bone turnover markers | 13 months
  Changes of C-terminal telopeptide of type I collagen (CTX) and propeptide of procollagen type I (P1NP)
clinical osteoporotic fracture | 1 year
  any incidence of clinical osteoporotic fracture

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Yunlin branch, Douliu, Yunlin County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
after application